CLINICAL TRIAL: NCT04615650
Title: Non-operative Versus Operative Treatment of Suprasyndesmotic Ankle Fractures: A Prospective, Multicentre, Randomised Controlled Trial
Brief Title: RCT Comparing Non-operative vs Operative Treatment of Suprasyndesmotic Ankle Fractures.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sykehuset Innlandet HF (Other)
Collaborators: Oslo University Hospital (Other); Vestre Viken Hospital Trust (Other); Ostfold Hospital Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 169307
Record Dates: First submitted 2020-10-28; First posted 2020-11-04 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Ankle Fractures
Keywords: ankle fractures; surgical treatment; conservative treatment; weight-bearing
MeSH Terms: conditions — Ankle Fractures | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Intervention Model Description: Randomised controlled multicentre trial
Who Masked: Outcomes Assessor
Masking Description: Data will be plotted into a database by an independent blinded data manager.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Surgical treatment (Active Comparator): Patients randomised to operative treatment will have their surgery performed by an orthopaedic surgeon or by orthopaedic trainees under the supervision of a consultant, when fit for surgery. The surgical technique and choice of implants will be decided by the surgeon in order to closely resemble everyday clinical practice. The syndesmosis must be reduced (closed or open) and fixed. Postoperatively, the patients will be treated with an ankle orthosis for six weeks with weight-bearing as tolerated.
  Interventions: Procedure: Surgical treatment
- Non-surgical treatment (Experimental): Patients randomised to non-operative treatment are treated with an ankle orthosis for six weeks with weight-bearing as tolerated. Other types of casts can be used if preferred by the treating orthopaedic surgeon, but the cast must allow full weight-bearing and must prevent equinus position.
  Interventions: Device: Ankle orthosis

INTERVENTIONS:
Procedure: Surgical treatment — Surgical treatment of suprasyndesmotic ankle fractures
  Arms: Surgical treatment
Device: Ankle orthosis — Non-surgical treatment of suprasyndesmotic ankle fractures
  Arms: Non-surgical treatment

SUMMARY:
Weight-bearing radiographs will be used to evaluate the stability of suprasyndesmotic ankle fractures. Patients with stable fractures will be randomised to operative or non-operative treatment.

DETAILED DESCRIPTION:
Suprasyndesmotic fractures (Weber type C) are historically treated operatively because of the assumption that the distal tibiofibular syndesmosis is ruptured, leading to joint instability (Lauge-Hansen 1950, Boden 1989).

However, the medial deltoid ligament may function as the main stabiliser of the ankle joint by preventing external rotation of the talus and therefore maintains the dynamic congruity (Michelson 2007). Due to the stabilising effect of the deltoid ligament, an increasing number of transsyndesmotic fractures (Weber type B) are treated non-operatively with excellent results and without the burden of complications that accompany surgery (Gougoulias 2017, Mittal 2017, Bauer 1985).

The aims of the present study are to test the stability of suprasyndesmotic ankle fractures on weight-bearing radiographs and to evaluate the effect of non-operative versus operative treatment of stable suprasyndesmotic fractures.

The patients will have a weight-bearing (at least 50% of body weight) standing radiograph for the evaluation of the stability of the fracture. Patients with a congruent ankle mortise (i.e., stable fracture) on weight-bearing radiographs will be randomised to either operative (ORIF, reference treatment) or non-operative treatment (cast). Patients in both groups are allowed full weight-bearing.

Patients with an incongruent ankle mortise (i.e., unstable fracture) will be treated operatively according to current clinical practice and included in a parallel observational cohort study. Patients who are unwilling to participate in the intervention study are also invited to participate in the observational cohort study.

ELIGIBILITY:
Inclusion Criteria:

* patients who present with a closed, isolated fibular fracture classified as suprasyndesmotic (Weber C) with a medial clear space of less than 7 mm in mortise view on primary radiographs.
* presentation less than 14 days after the injury.

Exclusion Criteria:

* previous fractures or ligamentous injury to the injured ankle.
* pathological fracture.
* diabetic neuropathy or other neuropathies.
* drug abuse.
* inability to consent and/or comply.
* inability to understand Norwegian language.
* inability to walk unaided prior to the fracture.
* patients with a concomitant tibial fracture requiring surgical treatment are excluded, but patients with undisplaced concomitant tibial fractures can be included.
* patients from outside the catchment area of the recruiting hospitals. However, they can be included if they are willing to undergo follow-up visits at one of the recruiting hospitals.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2020-12-28 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Olerud-Molander Ankle Score (OMAS) | The main statistical analysis of the primary outcome will be based on the two-year follow-up.
  The primary outcome measure is the Olerud-Molander Ankle Score (OMAS), which is a condition-specific, patient-reported measure of ankle-fracture symptoms. OMAS ranges from 0 to 100, with higher scores indicating better outcomes and fewer symptoms.

SECONDARY OUTCOMES:
Ankle pain | The main statistical analysis of the outcome will be based on the two-year follow-up.
  Ankle pain is measured by the Numeric Rating Scale (NRS), which is an 11-point numeric scale ranging from 0 ("no pain") to 10 ("worst pain imaginable").
Manchester-Oxford Foot Questionnaire (MOxFQ) | The main statistical analysis of the outcome will be based on the two-year follow-up.
  Ankle-related symptoms are, in addition to the OMAS questionnaire, measured by the Manchester-Oxford Foot Questionnaire (MOxFQ). The MOxFQ is a 16-item questionnaire consisting of three subscales: walking/standing (w/s) problems (seven items), pain (p) (five items), and issues related to social interaction (si) (four items). Patients score each question on a five-point Likert scale ranging from 0 to 4, with 4 representing the worst stage. Raw scores are converted to a numeric scale ranging from 0 to 100, with 100 denoting the most severe symptoms.
EuroQol questionnaire (EQ-5D) | The main statistical analysis of the outcome will be based on the two-year follow-up.
  Quality of life is measured by the EuroQol questionnaire (EQ-5D). EQ-5D is a validated generic health-related quality-of-life instrument. It consists of two parts: EQ-5D descriptive part and EQ-5D visual analogue scale. The descriptive part in-cludes five dimensions (mobility, self-care, usual activities, pain/discomfort, and anxie-ty/depression), each with three possible answers ("no problems", "some problems", and "major problems"). EQ-5D VAS is a visual analogue scale of self-related overall health, ranging from 0 (worst imaginable health state) to 100 (best imaginable health state).
Radiographic results | The main statistical analysis of the outcome will be based on the two-year follow-up.
  Radiographic results (fracture healing, joint congruency, syndesmotic reduction and post-traumatic arthritis) is assessed by plain radiographs and computed tomography (CT). Post-traumatic arthritis is graded on radiographs according to van Dijk et.al.
Range of motion | The main statistical analysis of the outcome will be based on the two-year follow-up.
  Range of motion of both ankles will be assessed by a physiotherapist or surgeon (who are not directly involved in the study) using a goniometer to measure active loaded dorsiflexion.
Adverse events | The main statistical analysis of the outcome will be based on the two-year follow-up.
  Adverse events, including deep vein thrombosis, nerve injury, wound infection and other complications occurring during the 24 months of follow-up are registered. Reoperations and crossover from non-operative to operative treatment are also registered.

CONTACTS AND LOCATIONS:
Overall Officials: Håvard Furunes, PhD, Principal Investigator — Sykehuset Innlandet HF
Locations (4):
- Norway (4):
  - Vestre Viken Hospital Trust, Bærums verk, Akershus
  - Østfold Hospital Trust, Fredrikstad, Akershus
  - Sykehuset Innlandet HF, Gjøvik, Innlandet
  - Oslo University Hospital, Oslo, Oslo County

IPD SHARING:
Plan to Share IPD: No
We have planned to use all the IPD only within the present study group.

REFERENCES:
- [Derived] Saatvedt O, Riiser M, Frihagen F, Figved W, Madsen JE, Molund M, Furunes H. Non-operative versus operative treatment of suprasyndesmotic ankle fractures: protocol for a prospective, multicentre, randomised controlled trial. BMJ Open. 2024 Jan 8;14(1):e075122. doi: 10.1136/bmjopen-2023-075122. PMID 38191245